CLINICAL TRIAL: NCT00949208
Title: Development of Applications of the Given® Diagnostic System and Evaluation of Their Performance
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: RD-30
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Healthy people

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: The study population will consist of healthy volunteers who fulfill all the inclusion criteria and do not meet any of the exclusion criteria.

SUMMARY:
The purpose of this study is to support the development of Given® Diagnostic System applications.

DETAILED DESCRIPTION:
This clinical study is designed to support the development of new generations of the Given® Diagnostic System and Agile™ Patency System that will accomplish better visualization, better diagnostic capabilities and will improve the system ease of use from the physician as well as patient's point of view.

*The PillCam™ Capsules Capsule endoscopy using the PillCam™ capsule (Given Imaging Limited, Yoqneam, Israel) represents the newest imaging modality of the gastrointestinal tract without the need for invasive techniques, sedation, or radiation exposure1-35. Initially cleared for marketing in August 2001 as an adjunctive modality, the FDA in 2003 cleared PillCam™ SB (previously called M2A) as a stand alone tool for detecting small bowel abnormalities in those patients who meet the device's indications.

The PillCam™ SB provides visualization of the entire small bowel mucosa and is presently purely a diagnostic test without therapeutic or biopsy potential.

Before capsule endoscopy, enteroscopy was one of the methods for examining the small bowel tract, but the diagnostic value of this test for a wide variety of specific lesions is low due to inability to reach the entire length of the small bowel.

Other endoscopic techniques include, Sonde enteroscopy, and intraoperative enteroscopy, but these are limited for several reasons including significant technical difficulties, length of procedures, potential risks, and frequently incomplete small bowel examination36-38. To date more than 400,000 PillCam™ SB capsules were ingested world wide. The Given® Diagnostic System (GDS) for Small Bowel is now the Gold standard.

Additional PillCam™ capsules were developed and are used for diagnosing the Esophagus as well as the Colon.

The PillCam™ ESO system received FDA clearance as well as the CE mark early 2005. To date, thousands of PillCam™ ESO capsules were ingested in both clinical trials and regular clinical setup worldwide with numerous published clinical studies39-45.

The PillCam™ COLON capsule received CE marking on October 15th, 2006 and is cleared for marketing in Europe. It is now pending FDA clearance. To date, several hundreds of PillCam™ COLON capsules were ingested in numerous pilot studies and ongoing multi-center studies in Europe and USA34-35.

*The Agile™ Patency System Small and large bowel strictures are present in a large spectrum of diseases and clinical situations such as adhesion related diseases, Crohn's disease, patients who are post abdominal radiation treatment and patients who have undergone abdominal surgery46. Knowledge of intestinal patency in such patients will aid the physician in assessment and treatment of the patients.

The current methods for identifying intestinal strictures primarily include small bowel follow through (SBFT), enteroclysis, computed tomography (CT) and enteroscopy but the diagnostic value of these tests is low. Advanced strictures are often missed and some of these methods include radiation and others are invasive.

The Agile™ Patency System is designed to aid the gastroenterologist in verifying the patency of the GI tract. The system is essentially based on small identification tags, which are detected by radio frequency (RFID) encapsulated in a disintegrating capsule. The RFID tags have been marketed for many years for veterinary use. In animals they are injected sub-dermally and are used for life-long identification, marking and tracking47.

Preliminary results demonstrate that the Agile System performs as intended48. Future developments of the unique technology which make up the Agile patency capsule will broaden its range of uses and applications beyond simple patency testing.

Agile ingestions are estimated in the excess of three thousand worldwide.

ELIGIBILITY:
Inclusion criteria

1. Subject's age is between 18-75 years.
2. Subject is healthy.
3. Subject agrees to sign the Informed Consent Form.

Exclusion criteria

1. Female subject is pregnant.
2. Subject is known or is suspected to suffer from intestinal obstruction (symptoms such as severe abdominal pain with accompanying nausea or vomiting).
3. Subject has a pacemaker or other implanted electro-medical device.
4. Subject has undergone certain prior abdominal surgery of the gastrointestinal tract, (other than uncomplicated appendectomy or uncomplicated cholecystectomy) such as small bowel or colonic resection. This will be evaluated by the PI.
5. Subject has any condition, which precludes compliance with study and/or device instructions, such as swallowing problems.
6. Subject suffers from life threatening conditions.
7. Subject is currently participating in another clinical study that may directly or indirectly affect the results of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of healthy volunteers who fulfill all the inclusion criteria and do not meet any of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1225 (Actual)
Dates: Start 2008-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Assessment of new or modified features of the GDS presently under development | Within 7 Days
Capsule transition time throughout the all GI tract segments & Improved visualization of the mucosa and sub-mucosal structures (mostly by capsule modification) | Within 7 days
Improved automatic pathology identification & bowel cleanliness - index score | Within 7 days
Accuracy of capsule localization & Pathology size determination | Within 7 days

SECONDARY OUTCOMES:
Identify and evaluate any additional features beneficial to GDS applications. | within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Chowers, Prof., Principal Investigator — Rambam Health Care Campus; Ari Bergwerk, Dr., Principal Investigator — Given Imaging
Locations (2):
- Israel (2):
  - Rambam - Medical center, Haifa
  - Given Imaging Ltd, Yoqneam